CLINICAL TRIAL: NCT05457868
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM) - Salbutamol vs Long-acting Muscarinic Antagonists
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019A010961-9
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Salbutamol: Exposure group
  Interventions: Drug: Salbutamol
- Long-acting muscarinic antagonists (LAMA): Reference group
  Interventions: Drug: LAMA

INTERVENTIONS:
Drug: Salbutamol — Salbutamol claim is used as the exposure group.
  Groups: Salbutamol
Drug: LAMA — Long-acting muscarinic antagonists (LAMA) - umeclidinium, aclidinium, tiotropium, glycopyrolate, glycopyrronium - claim is used as the reference group.
  Groups: Long-acting muscarinic antagonists (LAMA)

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1j53_NBnEVQik4Ps5a9pZOvuHm1mWHCRZ3DAvI0y8NO8/edit?usp=sharing or Appendix A (https://drive.google.com/file/d/1uC_G8TJ1ujoJbas1p1gFaYFzY7Hw7xMq/view?usp=sharing) for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability).

Inclusion Criteria:

* 1. Aged >/= 65 years on the index date
* 2. No prior use of Salbutamol and Long-acting Muscarinic Antagonists (LAMA) anytime prior to cohort entry date
* 3. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 4. At least two claims with COPD diagnosis measured 365 days prior to drug initiation

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior history of nursing home admission in the 365 days prior to the cohort entry date

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing Salbutamol versus Long-acting muscarinic antagonists (LAMAs). The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 124117 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Time to dementia onset | Through study completion (a median of 120 days)
  Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.

SECONDARY OUTCOMES:
Time to Alzheimer's disease onset | Through study completion (a median of 120 days)
  Time to Alzheimer's disease onset. Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT05457868/Prot_SAP_001.pdf